CLINICAL TRIAL: NCT06992479
Title: Efficacy of Nasal High-flow Oxygen Therapy Combined With Sequential Non-invasive Ventilation in Patients With Chronic Obstructive Pulmonary Disease Complicated With Type II Respiratory Failure
Brief Title: Efficacy of HFNC Combined With Sequential NIV in Patients With COPD Complicated With Type II Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Yanmei Gu, Head Nurse, Beijing YouAn Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL-2023-052-K
Record Dates: First submitted 2025-05-12; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Nasal High Flow Oxygen Therapy; Noninvasive Ventilation; Respiratory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC combined with sequential NIV therapy group (Experimental)
  Interventions: Device: high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation (NIV)
- NIV therapy group (Active Comparator)
  Interventions: Device: NIV routine treatment

INTERVENTIONS:
Device: high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation (NIV) — The control group was treated with NIV routine treatment. During non-invasive ventilation, patients in both the intervention group and the conventional group will receive NIV through a full mask or nasal mask using any of the existing ventilators in the hospital. Usually, the ventilator was set to the pressure support ventilation mode, and the inspiratory pressure was adjusted to the maximum tolerance to obtain the ideal body weight of 6 ~ 8mL / kg of exhaled tidal volume, and the PEEP was set at 3 ~ 5cmH2O. FiO2 in both groups was set to maintain 88% -92% peripheral blood oxygen saturation.
  The study group was treated with nasal high-flow oxygen therapy combined with sequential non-invasive ventilation. Patients will receive high-flow oxygen therapy ventilator during the day and in the morning and evening awake time (manufacturer: Hunan Mingkang Zhongjin Medical Technology Co., Ltd., registration number: Xiangji Zhuzhun 20192080049, model: OH60A) treatment. At night (from 10 p.m. to 6
  Arms: HFNC combined with sequential NIV therapy group
Device: NIV routine treatment — Usually, the ventilator was set to the pressure support ventilation mode, and the inspiratory pressure was adjusted to the maximum tolerance to obtain the ideal body weight of 6 ~ 8mL / kg of exhaled tidal volume, and the PEEP was set at 3 ~ 5cmH2O. FiO2 in both groups was set to maintain 88% -92% peripheral blood oxygen saturation.
  Arms: NIV therapy group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation (NIV) in patients with chronic obstructive pulmonary disease complicated with type II respiratory failure. The main questions it aims to answer are:

What is the effect of high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation on arterial blood gas indicators in patients with chronic obstructive pulmonary disease and type II respiratory failure? What is the effect of high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation on pulmonary ventilation function in patients with chronic obstructive pulmonary disease and type II respiratory failure? What is the effect of high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation on vital signs in patients with chronic obstructive pulmonary disease and type II respiratory failure? What is the effect of high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation on the quality of life of patients with chronic obstructive pulmonary disease and type II respiratory failure? What is the effect of high-flow nasal cannula oxygen therapy (HFNC) combined with sequential non-invasive ventilation on complications in patients with chronic obstructive pulmonary disease and type II respiratory failure?

Participants will:

Receive NIV through a full mask or nasal mask using any of the existing ventilators in the hospital Receive other standard treatments according to the latest GOLD guidelines The general data of patients, arterial blood gas index, pulmonary ventilation function, vital signs index, quality of life and complications before and after treatment were collected.

ELIGIBILITY:
Inclusion Criteria:

* All subjects included in the study met the diagnostic criteria for AECOPD in the Global Initiative for Chronic Obstructive Pulmonary Disease (2014 Update);
* Age > 18 years old;
* All patients met the diagnostic criteria for type II respiratory failure in the eighth edition of ' Internal Medicine ', that was, arterial blood PaO2 < 50mmHg;
* The patient was conscious, without myocardial infarction, acute stroke, severe liver and kidney dysfunction, severe coagulation dysfunction and other diseases;
* The patient did not have life-threatening hypoxemia and severe hemodynamic instability, and did not need tracheal intubation or tracheotomy;
* Patients can cooperate with pulmonary function tests.

Exclusion Criteria:

* Patients with pneumothorax, mediastinal emphysema or severe thoracic deformity;
* Patients with bronchial asthma, interstitial pneumonia and other diseases;
* Patients with coma and disturbance of consciousness;
* The upper respiratory tract or facial injury and facial deformity, can not wear a good nose (face) mask;
* Patients with septic shock or severe heart, kidney, liver and other diseases;
* Sputum and sticky, unable to expectoration or prone to aspiration caused by airway obstruction.
* Automatic discharge or transfer, or due to non-respiratory serious diseases (including non-invasive ventilator complications, non-invasive ventilation treatment ineffective need to be changed to invasive ventilation), termination of the study patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
arterial blood gas indexes | before and after 7 days of BiPAP treatment
the first second forced expiratory volume | before and after 7 days of BiPAP treatment
forced vital capacity | before and after 7 days of BiPAP treatment
FEV1 / FVC | before and after 7 days of BiPAP treatment
FEV1 / predicted value | before and after 7 days of BiPAP treatment
PEF / predicted value | before and after 7 days of BiPAP treatment
heart rate | before and after 7 days of BiPAP treatment
respiratory rate | before and after 7 days of BiPAP treatment
blood pressure | before and after 7 days of BiPAP treatment
Quality of life | before and after 7 days of BiPAP treatment
  SF-36 comprehensively summarized the quality of life of respondents from eight aspects: physiological function, physiological function, physical pain, general health status, energy, social function, emotional function and mental health. The score range is 0-100. The higher the score, the better the situation.
Complications | before and after 7 days of BiPAP treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing You'an Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No